CLINICAL TRIAL: NCT01587560
Title: A Comparison Between a Pyrocarbon and a CoCr Shoulder Resurfacing Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danderyd Hospital (Other)
Collaborators: Ascension Orthopedics, Inc. (Industry); Swedish Shoulder and Elbow Arthroplasty Register (Unknown); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Olof Skoldenberg, Director of research, Orthopedic dept., Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PyroTITAN DS
Record Dates: First submitted 2012-02-17; First posted 2012-04-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: Shoulder; Arthroplasty; Pyrocarbon; Randomized controlled trial; Shoulder resurfacing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyrocarbon (Active Comparator): Patients receiving a shoulder surface replacement implant made of pyrocarbon (the PyroTITAN Humeral resurfacing Arthroplasty)
  Interventions: Device: PyroTITAN, Ascension Orthopedics, Inc.; Device: TITAN, Ascension Orthopedics, Inc.
- CoCr (Active Comparator): Patients receiving a shoulder surface replacement implant made of Cobalt-Chrome(CoCR) (the TITAN Humeral Resurfacing Arthroplasty)
  Interventions: Device: PyroTITAN, Ascension Orthopedics, Inc.; Device: TITAN, Ascension Orthopedics, Inc.

INTERVENTIONS:
Device: PyroTITAN, Ascension Orthopedics, Inc. — All patients will be operated on with a shoulder resurfacing implant. In one arm of the study, the patients will receive an implant made of pyrocarbon. In the second arm, the patients will receive an implant made of Cobalt-Chrome. Aside from the materials, the implant are of the same design.
  Other Names: TITAN, Ascension Orthopedics, Inc.
Device: TITAN, Ascension Orthopedics, Inc.

SUMMARY:
The purpose of the study is to investigate fixation to bone and the clinical results following shoulder resurfacing arthroplasty. The study will compare results between an implant made of Cobalt-Chrome(CoCr) and an implant made in pyrocarbon.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary osteoarthritis of the shoulder
* Age 40-75 years
* Patient capable of giving informed consent
* Patient agrees to comply with the study plan

Exclusion Criteria:

* Destruction of the proximal humerus
* Insufficient bone stock
* Deficient rotator cuff or earlier failed surgery of the rotator cuff
* Large muscle defects or insufficient blood supply in the affected arm
* Neuromuscular disorders
* Infection, untreated malignancy or transmittable disease preventing the patient from fulfilling the study
* Patient unwilling to comply with study regulations
* Patient with earlier allergic reaction to pyrocarbon
* Patient with known metastatic disease
* Patient who has been treated with more than 10 mg corticosteroids (e.g. Prednisone) daily within 3 months from surgery.
* Patient participating in other clinical study
* Patient in need of glenoid replacement

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Fixation to bone as measured with radiostereometric analysis (RSA) | 24 months
  Early migration of the implants will be measured with RSA at 3, 6, 12 and 24 months.

SECONDARY OUTCOMES:
Clinical results after surgery as measured with EuroQol-5D(EQ-5D), American Shoulder and Elbow Surgeons Score(ASES), Constant score, and Western Ontario Osteoarthritis of the Shoulder index(WOOS) | 24-48 months
  Outcome after surgery will be evaluated using the above mentioned scores performed by and independent and blinded investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic department, Danderyd Hospital, Stockholm, Stockholm County, Sweden